CLINICAL TRIAL: NCT06660485
Title: Establishment of a Cohort for ConTinuous COronary CTA SCanning And PredicTive Analysis of Plaque Progression (TOCCATA)
Brief Title: Establishment of a Cohort for Continuous Coronary Artery CTA Scanning and Predictive Analysis of Plaque Progression
Acronym: TOCCATA
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Prof., West China Hospital
Other Study IDs: WestChinaH-CVD-007
Record Dates: First submitted 2024-10-14; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: CAD - Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Continuous CCTA Scanning Cohort

SUMMARY:
This research develops risk prediction models for coronary artery stenosis and vulnerable plaques. The coronary artery stenosis model aims to predict stenosis using multimodal deep learning by integrating text, structured numerical data, and imaging features, focusing on metrics like maximum and cumulative stenosis. The vulnerable plaque model seeks to identify early formation indicators, allowing for timely interventions to prevent plaque rupture, using similar data integration techniques. Additionally, a decision support system is created, comprising a patient database, risk prediction models, and a high-risk alert module. This system facilitates real-time notifications to healthcare providers when risk thresholds are exceeded, enabling personalized treatment planning and improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone multiple consecutive CCTA examinations.

Exclusion Criteria:

Patients who have undergone only a single CCTA examination. Patients whose CCTA image quality is poor and cannot be analyzed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone multiple consecutive CCTA examinations.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Coronary Stenosis (MAXS) | 2 year
  In 18 vascular segments, each segment is scored based on the degree of stenosis. The scoring criteria are as follows: no stenosis (0%) is scored as 0 points, mild stenosis (1%-24%) is scored as 1 point, moderate stenosis (25%-49%) is scored as 2 points, significant stenosis (50%-69%) is scored as 3 points, severe stenosis (70%-99%) is scored as 4 points, and total occlusion (100%) is scored as 5 points. MAXS represents the score of the single segment with the highest score among the 18 vascular segments.

SECONDARY OUTCOMES:
Cumulative Coronary Stenosis (SIS): | 2 year
  Each segment with a lesion among the 18 vascular segments is assigned a score of 1 point. If a segment does not have a lesion, it is scored as 0 points. The total score of SIS is the sum of the scores of all vascular segments with lesions.
Segment Involvement Score (SSS): | 2 year
  First, each lesion is scored based on its degree of stenosis, using the same scoring criteria as MAXS. Then, the scores of each lesion are accumulated based on their degree of stenosis (no stenosis is 0 points, mild stenosis is 1 point, moderate stenosis is 2 points, significant stenosis is 3 points, severe stenosis is 4 points, and total occlusion is 5 points). Finally, the scores of the 18 vascular segments are summed to obtain SSS.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Sichuan, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided